CLINICAL TRIAL: NCT07369362
Title: A Multicenter Randomized Controlled Non-Inferiority Trial Comparing SwimCount Harvester® to Standard Sperm Preparation Methods in IVF Cycles With PGT-A
Brief Title: To Investigate if the Harvester® Improves Sperm Motility and Blastocyst Utilization (the Percent of Fertilized Eggs That Develop to the Point That They Are Able to be Transferred) in IVF Cycles.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MotilityCount aps (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #20250195
Record Dates: First submitted 2026-01-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Infertility; Male Infertility; InVitro Fertilization; Aneuploidy Rate; Euploidy Rate
Keywords: SwimCount Harvester; Microfluidic sperm selection; Microfluidic sperm preparation; Density gradient centrifugation; Male factor infertility; Preimplantation genetic testing; Euploidy; Aneuploidy; blastocyst; blastocyst utilization; usable blastocyst; embryo; sperm motility; in vitro fertilization; prospective randomized controlled trial; operational efficiency
MeSH Terms: conditions — Infertility; Infertility, Male; Aneuploidy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control group; standard sperm preparation and selection (No Intervention): This arm is the control group and patients randomized to this arm of the study will have semen processed according to standard operating procedures.
- Study group - microfluidics device for sperm preparation (Experimental): Patients randomized to this arm will have their semen processed using the SpermHarvest device which is an FDA approved microfluidics device for semen processing.
  Interventions: Device: microfludics semen processing device

INTERVENTIONS:
Device: microfludics semen processing device — Semen will be processed through this device for patients randomized to the study group arm. It is the only intervention.
  Arms: Study group - microfluidics device for sperm preparation

SUMMARY:
The goal of this prospective, multicenter randomized controlled clinical trial is to evaluate whether the SwimCount Harvester microfluidic sperm preparation device can achieve equivalent or superior clinical outcomes compared to standard sperm preparation methods (density gradient centrifugation and swim-up) in couples undergoing in vitro fertilization (IVF) with preimplantation genetic testing for aneuploidy (PGT-A).

The study population includes adult couples (female partner age 21-45 years; male partner age ≥21 years) undergoing IVF with PGT-A who meet minimum semen eligibility criteria on the day of oocyte retrieval: pre-processing volume ≥1mL, sperm concentration ≥1 million/mL, and progressive motility ≥10%. A total of 1,600 patients will be randomized 1:1 across 15-25 high-volume IVF centers to receive either Harvester or the site's predominant standard-of-care sperm preparation method. Patients with surgical sperm retrieval requirements or those currently using SwimCount Harvester as standard of care are excluded.

The main questions it aims to answer are:

Does the SwimCount Harvester demonstrate noninferiority to standard sperm preparation methods on blastocyst utilization rate? The primary endpoint is blastocyst utilization rate, calculated as the number of usable blastocysts (operationalized as biopsied blastocysts per clinic standard operating procedures) divided by the number of normally fertilized oocytes (2PN) at the patient level. Noninferiority will be concluded if the lower bound of the two-sided 95% confidence interval for the risk difference (Harvester minus standard of care) is greater than -2.0 percentage points, using a site-stratified Mantel-Haenszel analysis. If noninferiority is met, superiority may be reported as supportive evidence when the lower confidence bound exceeds zero.

Does the SwimCount Harvester demonstrate noninferiority to standard sperm preparation methods on the probability of obtaining at least one euploid embryo per retrieval? The key secondary endpoint assesses whether patients have at least one euploid embryo (yes/no) based on PGT-A results from a single blinded reference laboratory (NOVA Genomics). This will be analyzed as a site-stratified Mantel-Haenszel risk difference with a two-sided 95% confidence interval, with an optional noninferiority margin of -2.5 percentage points presented as supportive evidence.

Additional supportive and exploratory questions include:

* How does progressive motility change from pre- to post-preparation with each method? Progressive motility will be summarized descriptively pre- and post-preparation as a supportive laboratory measure without hypothesis testing.
* Do outcomes differ in clinically important subgroups? Pre-specified exploratory analyses will examine advanced maternal age (≥40 years) and severe oligospermia (<5 million/mL), populations that may derive differential benefit from advanced sperm selection.
* What are the practical implementation considerations? An independent protocol complexity analysis will assess procedural steps, equipment requirements, and standardization benefits by comparing site standard-of-care protocols to the Harvester Instructions for Use.

The study addresses a critical evidence gap by providing multicenter, adequately powered data on whether advanced microfluidic sperm preparation translates into meaningful clinical improvements in IVF success metrics.

DETAILED DESCRIPTION:
DETAILED DESCRIPTION Scientific Background and Rationale Infertility affects 10-15% of couples globally, with male factors contributing to nearly half of cases. Sperm preparation is a critical laboratory step in assisted reproductive technology (ART) that directly influences clinical outcomes beyond baseline semen quality. Density gradient centrifugation (DGC) and swim-up have been the prevailing sperm preparation techniques for decades, but both methods are labor-intensive, require multiple procedural steps, and can generate inter-laboratory variation due to technique-dependent factors.

DNA Fragmentation and Sperm Selection The clinical advantage of modern sperm separation techniques stems from reductions in sperm DNA fragmentation. Meta-analyses of microfluidic sperm selection demonstrate significant improvements in DNA fragmentation (mean difference -9.98%, p<0.00001), progressive motility (mean difference +14.50%, p=0.04), and fertilization rates (OR 1.22, p=0.04). Crucially, these gains are independent of baseline semen metrics, suggesting that preparation method choice can compensate for poor starting material-particularly relevant for severe oligospermia populations.

Progressive Motility as a Surrogate Biomarker Progressive motility serves as more than a functional measure; it acts as a surrogate for sperm genomic integrity and predicts embryo developmental trajectory. High-motility sperm reliably exhibit lower DNA fragmentation, superior chromatin organization, and optimized mitochondrial function. Published evidence demonstrates that higher post-preparation progressive motility significantly enhances blastocyst formation rates in ICSI cycles (42.7% vs 28.2%, p=0.015), and motility correlates closely with fertilization (p=0.012), pregnancy (p=0.001), and live birth rates (p=0.001) in IVF.

Severe Oligospermia as a Distinct Clinical Challenge Multicenter studies demonstrate that men with severe oligospermia (<5 million/mL) face 12-15% lower fertilization and 18-22% lower blastulation rates, even after adjustment for female age and other variables. Their sperm also exhibit worse DNA fragmentation and chromatin quality, creating a distinct pathophysiological state that may derive differential benefit from advanced sperm selection technologies.

Study Design and Methodology Trial Architecture This is a prospective, multicenter, randomized (1:1), parallel-arm, noninferiority trial with PGT-A laboratory blinding. The trial compares the SwimCount Harvester microfluidic sperm preparation device to each site's predominant standard-of-care method across 15-25 high-volume IVF centers. Sites where DGC or swim-up constitute ≥90% of standard practice will comprise the primary analysis cohort; sites already using microfluidic devices as standard of care will be analyzed exploratorily to capture real-world diversity.

Device Description and Mechanism The SwimCount Harvester (MotilityCount ApS, Copenhagen, Denmark) is an FDA 510(k)-cleared (K241348, January 2025) and CE-marked (EU MDR 2017/745) Class II medical device for sperm preparation in assisted reproduction. The device employs micro-scale, membrane-mediated motility selection: motile sperm traverse a microporous barrier from the sample reservoir to a harvest compartment during 30-60 minute incubation at 37°C. This passive selection process isolates sperm with higher progressive motility and lower DNA fragmentation without the mechanical stress of centrifugation. Available in 1 mL and 3 mL cartridges, the device is single-use and requires minimal technical training (1-2 hours).

Randomization and Allocation Participants are randomized on the day of oocyte retrieval after eligibility confirmation and pre-preparation semen analysis (volume, concentration, progressive motility). Randomization uses permuted variable-size blocks within site, with 1:1 allocation to Harvester or site standard of care. Allocation concealment is maintained via the Sealed Envelope electronic system (ISO/IEC 27001 certified, 21 CFR Part 11 compliant), which reveals only the next assignment at the time of randomization.

The electronic data capture (EDC) system gates randomization based on real-time eligibility verification: semen volume ≥1mL, concentration ≥1 million/mL, progressive motility ≥10%, and signed informed consent on file. If any criterion is unmet, randomization is not released and the cycle is recorded as a screen failure.

Blinding Strategy Embryologists performing sperm preparation cannot be blinded due to the visible differences between devices and methods. However, critical outcome assessments are protected from bias: all PGT-A analyses are performed by a single reference laboratory (NOVA Genomics, Provo, UT) blinded to treatment arm assignment. Embryo grading is performed by site embryologists according to their established standard operating procedures without central grading, preserving real-world external validity. The blinded PGT-A laboratory reports euploidy, aneuploidy, and mosaic status using standardized criteria.

Site Selection and Method Distribution Sites must perform ≥200 IVF cycles with PGT-A annually and maintain a predominant sperm preparation method in ≥90% of cases. Target method distribution: 70% of sites using DGC/swim-up as standard of care (primary analysis cohort) and up to 30% using microfluidic devices as standard of care (exploratory cohort). A patient-weight safeguard ensures that ≥75% of control-arm patients are prepared with DGC/swim-up to maintain statistical power for the primary comparison. Quarterly monitoring reviews assess method distribution; if microfluidic standard-of-care enrollment exceeds 25% of control patients, a blinded power assessment (using observed baseline rates without treatment-effect unblinding) will determine whether enrollment restrictions are needed.

Laboratory Standardization

To minimize inter-site variability, each participating site must:

* Use the same culture media formulation across all enrolled patients regardless of randomization arm
* Use the same sperm counting method (manual vs CASA) and chamber type across all enrolled patients
* Use the same counting method and timing for both pre- and post-preparation progressive motility assessments
* Maintain these methods unchanged throughout the study period Temperature handling differs by design to reflect real-world practice: the Harvester arm follows the device instructions for use (37°C incubation), while the standard-of-care arm follows each site's validated standard operating procedure. These differences are not considered protocol deviations.

Data Collection and Management Streamlined Data Capture To minimize site burden while capturing high-quality data, the protocol employs a minimal case report form (CRF) requiring <2 minutes per cycle for essential fields: patient ID, site identifier, treatment arm, 2PN count, usable blastocyst count, pre-preparation progressive motility, and post-preparation progressive motility. Optional metadata (blastocyst day of development, Gardner grade, DNA fragmentation, morphology) are collected when available but do not delay enrollment.

Technology Integration Where available, Alife Health's Embryo Assist software integrates seamlessly with existing microscope hardware, allowing embryologists to capture embryo images and enter data in a centralized location without workflow disruption. Sites without Embryo Assist installation may proceed using the minimal CRF alone; image capture is optional and will not delay enrollment. This no-stall implementation strategy ensures that technology adoption does not impede recruitment timelines.

Device Tracking and Quality Assurance All SwimCount Harvester cartridges are tracked via lot number documentation in the CRF to ensure traceability and support quality assurance. Devices are provided in-kind by the sponsor (MotilityCount ApS) with no monetary compensation to sites or investigators. Device deficiencies (e.g., membrane clogging, which occurs in <1% of uses per manufacturer data) are documented as adverse events and reported to the sponsor and FDA as required.

Endpoint Definitions The primary endpoint-blastocyst utilization rate-is calculated as the number of usable blastocysts divided by the number of normally fertilized oocytes (2PN) at the patient level. Because all cycles in this study undergo PGT-A, "usable blastocysts" are operationalized as blastocysts biopsied for genetic testing per clinic standard operating procedures. This definition ensures consistency across sites while reflecting the clinical decision to biopsy an embryo deemed suitable for potential use.

The key secondary endpoint-probability of at least one euploid embryo per retrieval-is a binary (yes/no) outcome based on PGT-A results from the blinded central laboratory. This patient-centered measure directly assesses whether the intervention increases the likelihood of having a transferable euploid embryo.

Progressive motility is summarized descriptively (pre- and post-preparation, with change scores) as a supportive laboratory measure without hypothesis testing. Additional exploratory endpoints include counts and proportions of euploid vs aneuploid embryos, risk of having zero usable blastocysts per cycle, and optional DNA fragmentation and morphology assessments.

Statistical Analysis Approach Primary Estimand and Decision Rule The primary estimand is the risk difference in blastocyst utilization rate (Harvester minus standard of care) at the patient level in the index cycle, analyzed in the intent-to-treat population (all randomized patients). The analysis employs a site-stratified Mantel-Haenszel risk difference with a two-sided 95% confidence interval. Noninferiority is concluded if the lower confidence bound exceeds -2.0 percentage points. If noninferiority is met, superiority may be reported when the lower confidence bound exceeds zero; this superiority statement is supportive and does not alter the primary conclusion.

Noninferiority Margin Justification

The -2.0 percentage point noninferiority margin for blastocyst utilization was selected based on:

1. Clinical relevance: the margin corresponds to approximately 10-15% of typical inter-site natural variation observed in site audits (observed range: 12-18 percentage points across high-quality IVF centers)
2. Preservation of standard-of-care performance: the margin preserves ≥90% of control-arm performance
3. Regulatory guidance: the margin aligns with ICH E10 principles for noninferiority trial design
4. Patient impact: mapping the margin to patient-centered outcomes (e.g., probability of ≥1 euploid embryo) shows an expected absolute impact ≤3 percentage points, which is clinically negligible Sample Size and Power With 800 patients per arm across ≥15 sites, the study has ≥80% power to demonstrate noninferiority at the -2.0 percentage point margin when the true difference is between 0 and +5 percentage points and the standard-of-care blastocyst utilization rate is approximately 50%. If the true difference is +7 percentage points (50% to 57%), the study has approximately 80% power to demonstrate superiority at two-sided alpha=0.05.

For the key secondary endpoint (≥1 euploid embryo per retrieval), assuming a baseline rate of 45% in the standard-of-care arm, 800 patients per arm provides approximately 80% power to demonstrate noninferiority at a -2.5 percentage point margin when the true difference is between 0 and +5 percentage points.

The Mantel-Haenszel stratified analysis accounts for site-level clustering by stratifying on site. Power calculations assume a low intraclass correlation coefficient (ICC=0.03) based on observed inter-site homogeneity in contemporary PGT-A freeze-all protocols across participating centers. Baseline rates (50% blastocyst utilization, 45% probability of ≥1 euploid embryo) were validated against pre-study site audits and contemporary multicenter observational data.

Handling of Missing Data and Zero Fertilization For the primary endpoint, if both numerator (usable blastocysts) and denominator (2PN) are missing, blastocyst utilization is conservatively set to 0%. Sensitivity analyses include: (i) complete-case analysis and (ii) excluding cycles with missing blastocyst utilization data.

For cycles with zero fertilization (2PN=0), blastocyst utilization is set to 0% in the primary intent-to-treat analysis, reflecting treatment failure. A sensitivity analysis excludes zero-fertilization cycles to assess robustness.

For the key secondary endpoint, if euploidy status is missing, the patient is conservatively treated as having no euploid embryo; a complete-case sensitivity analysis will be reported.

If either pre- or post-preparation progressive motility is missing, the change score is missing and that patient is excluded from progressive motility summaries (complete-case only).

Quality standards target ≤5% patient-level missingness for primary endpoints and ≤10% for secondary endpoints.

Multiplicity Control There is one primary endpoint (blastocyst utilization rate) with a single noninferiority test; no multiplicity adjustment is required. The key secondary endpoint (≥1 euploid embryo) is analyzed inferentially but does not affect the primary conclusion; results are interpreted as supportive evidence. All other secondary and exploratory endpoints are analyzed without adjustment for multiple comparisons, with results interpreted as exploratory and hypothesis-generating.

Subgroup Analyses

Pre-specified subgroup analyses include:

1. Advanced maternal age (≥40 years): expected n=320 patients (20% of cohort)
2. Severe oligospermia (<5 million/mL): analyzed exploratorily based on evidence that this population experiences significantly compromised ICSI outcomes despite bypass of natural selection barriers, suggesting advanced sperm selection may provide disproportionate benefit
3. Standard preparation method: DGC vs swim-up within conventional standard-of-care sites (primary analysis); microfluidic standard-of-care sites analyzed separately (exploratory) Subgroup effects will be reported with 95% confidence intervals when N≥100 per arm within the subgroup; otherwise, results will be descriptive only. No interaction p-values will be calculated to avoid false-positive findings in underpowered comparisons.

Interim Monitoring There will be no formal interim efficacy or futility analysis. A single interim review at approximately 50% of planned information (defined as the point when both 2PN and blastocyst utilization data are available for 50% of target cycles) will assess safety, data quality, and operational progress only, without treatment-effect unblinding.

Protocol Complexity and Workflow Efficiency Analysis

Beyond clinical endpoints, the study includes a unique protocol complexity analysis to inform real-world implementation decisions. The independent study team will review all submitted site standard-of-care protocols and the SwimCount Harvester Instructions for Use to assess:

* Number of procedural steps required
* Equipment and consumable requirements
* Technical skill requirements and training burden
* Protocol standardization potential across sites Method-specific summaries for DGC, swim-up, and microfluidic methods will support laboratory adoption decisions. No site-level timing data will be collected; the analysis is based solely on protocol documents submitted at study initiation. This approach directly addresses laboratory directors' primary concerns regarding implementation feasibility without adding site burden.

Safety Monitoring The SwimCount Harvester is an FDA 510(k)-cleared and CE-marked medical device with an established safety profile. The study involves no invasive procedures beyond routine IVF sperm preparation, limiting physical risks to those inherent in standard DGC or swim-up methods (e.g., minor exposure to centrifugation media). No additional physical hazards are introduced by the microfluidic Harvester device.

Adverse events and device deficiencies will be documented and reported per standard clinical trial procedures to the IRB and sponsor. Serious adverse events (SAEs)-defined as any event requiring medical intervention beyond routine IVF care-will be reported within 24 hours to the IRB and sponsor, with non-serious AEs reported at routine monitoring intervals. Device-related AEs include any device malfunction requiring use of a backup preparation method.

Given the device's cleared status and established safety profile, no independent Data and Safety Monitoring Board is required. An independent monitor will review safety data at the interim operational checkpoint to determine whether unforeseen issues warrant study modification or halting, though none are anticipated given the device's low-risk classification.

Regulatory and Ethical Considerations Informed Consent Informed consent is obtained from both partners at least 24 hours prior to oocyte retrieval to allow adequate time for consideration and questions. Randomization occurs on the day of retrieval after confirming continued participation and verifying eligibility criteria. Participants may withdraw at any point without affecting their clinical care.

Conflicts of Interest This study is sponsored by MotilityCount ApS, the manufacturer of the SwimCount Harvester device. The sponsor provides in-kind support through donation of study devices (1 mL and 3 mL cartridges) and training for participating sites, valued at approximately $50,000 based on site projections. No monetary compensation, financial incentives, payments, or equity interests are provided to principal investigators, site staff, or participants.

Data management and randomization are provided by Sealed Envelope Ltd., a contracted service provider with no financial interest in study outcomes. Statistical analysis is conducted independently by a study statistician with no financial relationship with MotilityCount ApS. The central PGT-A laboratory (NOVA Genomics) has no knowledge of treatment arm assignments and no financial interest in study outcomes.

IRB Review and GCP Compliance The study will be reviewed by a Central IRB (WCG Clinical) with participating sites operating under reliance agreements where permitted by institutional policy. The lead Principal Investigator holds current CITI GCP (FDA Devices) and CITI Biomedical/Behavioral Investigator and Social & Behavioral Research certifications and is solely responsible for ensuring GCP compliance across all sites. Site personnel will receive study-specific GCP training via a 30-60 minute virtual session conducted by the lead PI or designee, covering protocol adherence, informed consent, adverse event reporting, data integrity, and delegation. No independent CITI certification is required for site staff; meeting documentation and attestation forms signed post-session confirm understanding.

Data Privacy and Protection Data are de-identified and managed in compliance with HIPAA (U.S. sites) and GDPR (EU sites). The EDC system (Sealed Envelope Red Pill) is 21 CFR Part 11 compliant and GCP validated. Cross-border data transfers will use standard contractual clauses or equivalent safeguards where applicable.

With participant consent, de-identified data may be retained in a sponsor-managed research repository for up to 15 years and used for future IRB/EC-approved studies related to assisted reproduction, laboratory workflow, and embryo assessment methods. External access (academic or commercial) will require a Data Use Agreement and approval by the study Data Access Committee. Participants may withdraw consent for future use at any time prior to de-identification.

Secondary and Exploratory Analyses

The study dataset may be made available for pre-specified secondary analyses following completion of the primary study and publication of primary results. Anticipated secondary analyses include:

1. AI Algorithm Validation: Analysis of embryo morphology data captured via Embryo Assist to validate AI-based prediction models for embryo euploidy, in collaboration with Alife Health. This analysis will correlate morphology assessments, time-lapse parameters, and euploidy outcomes to improve predictive algorithms for embryo developmental potential and genetic competence.
2. Subgroup and Method-Specific Analyses: Additional analyses of workflow efficiency by patient subgroups, correlation analyses between sperm parameters and downstream embryo outcomes, and preparation method-specific effectiveness analyses.
3. Meta-Analysis Contribution: Anonymized individual patient data may be contributed to systematic reviews and meta-analyses examining sperm preparation techniques in ART to enhance evidence synthesis.

All secondary analyses will use fully anonymized datasets with patient identifiers removed per HIPAA Safe Harbor standards. Secondary analyses require separate IRB approval or exempt determination prior to initiation. AI algorithm development will comply with institutional AI governance policies and FDA guidance on AI/ML in medical devices.

Study Timeline

* Months 0-1: Site qualification, selection, contracting; Sealed Envelope EDC/randomization system setup; Embryo Assist software preparation
* Month 2: Site training, IRB approvals, Embryo Assist installation and validation
* Months 3-16: Patient enrollment (target: 115 patients/month across all sites)
* Month 17: Database lock and preliminary analysis
* Month 18: Complete statistical analysis and quality checks
* Month 19: Final statistical report
* Month 20: Manuscript preparation and conference abstracts Total enrollment period: 14 months (Months 3-16). Expected Impact This study addresses a critical evidence gap in reproductive medicine by providing the first adequately powered, multicenter randomized controlled trial to determine whether advanced microfluidic sperm preparation translates into meaningful improvements in clinical IVF outcomes. Existing studies are limited by small sample sizes, single-center designs, and inconsistent comparator arms, with a striking lack of method-specific analyses or power for subgroup exploration.

An anticipated gain of 7.0 percentage points in blastocyst utilization could reduce the number of IVF cycles needed per live birth, advancing care for millions of couples affected by male factor infertility. Progressive motility improvements (expected +7.5 percentage points) will be assessed as supportive laboratory measures of sperm quality enhancement.

By combining rigorous clinical endpoint assessment with practical workflow analysis, this trial will empower ART laboratories with high-quality evidence for sperm preparation method selection, supporting precision medicine approaches in reproductive care.

ELIGIBILITY:
Inclusion Criteria:

* • Sperm sample available on day of egg retrieval

  * Female partner age 21-45 years undergoing IVF with PGT-A
  * Male partner age ≥ 21 years
  * Pre-processing volume ≥1mL
  * Pre-processing sperm concentration ≥1 million/mL
  * Pre-processing progressive motility ≥10%
  * Signed informed consent from both partners

Exclusion Criteria:

* • Surgical sperm retrieval required

  * Current standard of care with the SwimCount Harvester device

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1600 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Useable Blastocyst Rate | One week - from the day of oocyte retrieval through the last day of embryo assessment.
  Percentage of blastocysts cryopreserved per number of fertilized oocytes.

SECONDARY OUTCOMES:
Number of euploid blasts per cycle | From the start of an IVF cycle through its completion at 15-28 days.
  The number of blastocysts that have a normal PGT result per cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- First Fertility, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie results in published manuscripts will be made available to qualified researchers following publication of primary study results. The dataset will include demographics, sperm parameters (pre- and post-preparation concentration, progressive motility), blastocyst utilization data (2PN count, usable blastocyst count), PGT-A results (euploidy status), and randomization assignment. Optional variables collected when available include DNA fragmentation, sperm morphology, blastocyst development day, and Gardner grade. Data will be irreversibly de-identified per HIPAA Safe Harbor standards before sharing. Requests must include a methodologically sound proposal with scientific aims related to assisted reproduction, laboratory workflow, or embryo assessment methods.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: at the conclusion of the study

REFERENCES:
- [Background] Donnelly ET, Lewis SE, McNally JA, Thompson W. In vitro fertilization and pregnancy rates: the influence of sperm motility and morphology on IVF outcome. Fertil Steril. 1998 Aug;70(2):305-14. doi: 10.1016/s0015-0282(98)00146-0. PMID 9696226
- [Background] Gisbert Iranzo A, Cano-Extremera M, Hervas I, Falquet Guillem M, Gil Julia M, Navarro-Gomezlechon A, Pacheco-Rendon RM, Garrido N. Sperm Selection Using Microfluidic Techniques Significantly Decreases Sperm DNA Fragmentation (SDF), Enhancing Reproductive Outcomes: A Systematic Review and Meta-Analysis. Biology (Basel). 2025 Jun 30;14(7):792. doi: 10.3390/biology14070792. PMID 40723352
- [Background] Nosrati R, Vollmer M, Eamer L, San Gabriel MC, Zeidan K, Zini A, Sinton D. Rapid selection of sperm with high DNA integrity. Lab Chip. 2014 Mar 21;14(6):1142-50. doi: 10.1039/c3lc51254a. PMID 24464038
- [Background] Quinn MM, Jalalian L, Ribeiro S, Ona K, Demirci U, Cedars MI, Rosen MP. Microfluidic sorting selects sperm for clinical use with reduced DNA damage compared to density gradient centrifugation with swim-up in split semen samples. Hum Reprod. 2018 Aug 1;33(8):1388-1393. doi: 10.1093/humrep/dey239. PMID 30007319
- [Background] Bartolacci A, Pagliardini L, Makieva S, Salonia A, Papaleo E, Vigano P. Abnormal sperm concentration and motility as well as advanced paternal age compromise early embryonic development but not pregnancy outcomes: a retrospective study of 1266 ICSI cycles. J Assist Reprod Genet. 2018 Oct;35(10):1897-1903. doi: 10.1007/s10815-018-1256-8. Epub 2018 Jul 11. PMID 29995229